CLINICAL TRIAL: NCT04082052
Title: Evaluating and Predicting Response to a Single Session Intervention for Self-Dislike
Acronym: GOALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB2019-00312
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Depressive Symptoms; Self-Appraisal
Keywords: depression; self-dislike; self-compassion; symptom level; single session
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants will be randomized by Qualtrics and will be unknown to the investigator and the patient until data collection is complete
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Session Intervention for Self-Dislike (Experimental): A 30-45 minute intervention delivered in a web browser that focuses on reducing self-dislike using facts about the brain, testimonials from peers, and writing exercises.
  Interventions: Behavioral: Single Session Interventions
- Single Session Intervention for Feelings Disclosure (Placebo Comparator): A 30-45 minute intervention delivered in a web browser that focuses on encouraging feelings disclosure using facts about the brain, testimonials from peers, and writing exercises.
  Interventions: Behavioral: Single Session Interventions

INTERVENTIONS:
Behavioral: Single Session Interventions — A single session intervention either active (for self-dislike) or placebo (feelings disclosure)

SUMMARY:
The investigators are testing whether a single session online intervention for self-dislike decreases:

1. Fear of self-compassion from immediate pre to immediate post intervention
2. Self-hatred immediate pre to 1 month post-intervention
3. Individual depression symptoms immediate pre to 1 month post-intervention more than a placebo online single session intervention encouraging the disclosure of feelings in college students.

   The investigators will also explicitly test whether the following variables are predictors, of at least the smallest variance predicted of interest, of response to treatment vs. placebo on self-hatred:
4. Pre intervention self-hatred score
5. Screening positive for clinical depression based on self-report
6. Immediate pre to post-intervention reduction in fear of self-compassion
7. The investigators will also assess whether any of the variance shared between the treatment and changes in individual depression symptoms immediately pre Intervention to 1 month post-intervention is statistically mediated by change in self-hatred from immediate pre intervention to 1 month post intervention

ELIGIBILITY:
Inclusion Criteria:

Participant is a current college student at the time of study enrollment

Participant has not previously taken part in the study

Participant speaks English well enough to complete online intervention activities, which are available in English only

Participant is comfortable with completing online surveys and programs

Participant is at least 18 years of age.

Exclusion Criteria:

The investigators will exclude participants 3 SDs above/below the mean completion time for the study or exit the study prior to randomization for our listed analyses.

The investigators will also test whether there's any association between how quickly participants are responding to questions and the variability in their responses. If there is a response time frame (i.e., a series of questions that require answers where timing is measured) where there is a linear relationship between response time and response variability, the investigators may exclude those participants, as response time and response variability should be uncorrelated and a linear association can indicate random responding. This time frame can be identified visually on a graph, and sensitivity tests can be conducted to determine if slight variations on the visual interpretation affect substantive results.

The investigators will exclude participants who respond with either copy/pasted responses from text earlier in the intervention (e.g. Copy and pasting only text from a previous testimonial slide) to any of free response questions.

The investigators will exclude for primary analyses (but may run sensitivity analyses including them) any participants who provide responses of 5 words or fewer to writing prompts that ask for at least 1 sentence or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fear of Self-Compassion by Condition | Immediate pre intervention to 0-2 minute follow up post-intervention
  Self-report average score from the fear of self-compassion scale. Participants rate 15 items on a scale reflecting different fears/barriers to being self-compassionate they experience. Average scores range from 1-5. Higher scores indicate a greater fear of self-compassion.
Change in Self-Hatred by Condition | Immediate pre intervention to one month follow-up
  Self-report average score from the self-hatred scale. Participants rate 7 items on a scale reflecting their levels of self-dislike/self-hatred. Average scores range from 1-7. Higher scores indicate a greater self-hatred.
Change in Individual Depressive Symptoms by Condition | Immediate pre intervention to one month follow-up
  Self-report average score from the individual symptoms on the IDAS-II Dysphoria scale. Participants rate 10 items on a scale reflecting their experience of depression symptoms that all load onto one latent factor. Average scores range from 1-5. Higher scores indicate experiencing more of a given symptom.

SECONDARY OUTCOMES:
Change in Verbally Expressed Emotion-Sadness | Immediate pre intervention to 0-2 minute follow up post-intervention
  Self-report average score of verbally expressed emotion-sadness scale. Participants rate 3 items reflecting their willingness to disclose sadness to others. Average scores range from 1-4. Higher scores indicate less willingness to disclose sadness to others.
Change in PHQ-9 Depression Symptoms | Immediate pre intervention to one month follow-up
  Self-report average score of depression symptoms on the PHQ-9 scale. Participants rate 9 items related to depression symptoms they've experienced in the past two weeks. Average scores range from 0-3. Higher scores indicate more depression symptoms
Change in the Self-Dislike Item of the BDI-II Depression Symptom | Immediate pre intervention to one month follow-up
  Self-report score of the BDI II Self-Dislike item. Participants rate 1 item related to self-dislike on a scale from 0-3. A higher score indicates more self-dislike.
Change in Drinking to Cope Scale | Immediate pre intervention to one month follow-up
  Self-report average score of the Drinking to Cope scale. Participants rate 5 items on how often they drink alcohol to cope with difficulties. Average scores range from 1-5. Higher scores indicate greater frequency in drinking to cope.
Change in Social Phobia Screener | Immediate pre intervention to one month follow-up
  Self-report average score of the Social Phobia Screener scale. Participants rate 5 items on how socially anxious they have been in the previous month. Average scores range from 0-4. Higher scores indicate more social anxiety
Change in Brief Emotional Intelligence Scale | Immediate pre intervention to one month follow-up
  Self-report average score of the Brief Emotional Intelligence scale. Participants rate 10 items reflecting their self-perceived emotional intelligence. Average scores range from 1-5. Higher scores indicate greater self-perceived emotional intelligence.
Change in Empathy | Immediate pre intervention to one month follow-up
  Self-report average score of the Mutual Psychological Development scale. Participants rate 22 items on how often they reacted in certain ways in the past ways when talking with others about things that mattered to them. Average scores range from 1-6. Higher scores indicate greater empathy.
Understanding of the Intervention: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how much the participant understood the intervention. Participants rate 1 item on a scale from 1 to 5 on how well they understood the intervention. Higher scores indicate greater self-reported understanding of the intervention.
Effort Put Into the Intervention: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how much self-reported effort the participant put into the intervention. Participants rate 1 item on a scale from 1 to 5 on how much effort they put into completing the intervention. Higher scores indicate greater self-reported effort put into the intervention.
Interest in the Intervention: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how much self-reported interest the participant had about the intervention. Participants rate 1 item on a scale from 1 to 5 on how much interest they had in the intervention. Higher scores indicate greater self-reported interest in the intervention.
Perceived Logicalness of the Intervention: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how logical the participant believed the intervention to be. Participants rate 1 item on a scale from 1 to 9 on how logical they believed the intervention to be. Higher scores indicate greater self-reported logicalness in the intervention.
Confidence in Recommending the Intervention to a Friend: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how confident the participant would be in recommending the intervention to a friend who was struggling. Participants rate 1 item on a scale from 1 to 9 on how confident they would be in recommending these materials to a friend. Higher scores indicate greater self-reported confidence in recommending the intervention to a friend who was struggling.
Confidence in the Intervention Material's Ability to Improve Emotional Difficulties: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how confident the participant is that the intervention will help improve their own emotional difficulties. Participants rate 1 item on a scale from 1 to 7 on how confident they are the intervention materials will improve their emotional difficulties. Higher scores indicate greater self-reported confidence that the intervention materials would improve their own emotional difficulties.
Relevance to College Student's Lives: Self-report | 0-2 minute follow up post-intervention
  Self-report score on how relevant the intervention is to college students. Participants rate 1 item on a scale from 1 to 7 on how relevant the intervention materials are to college students. Higher scores indicate greater self-reported relevance of the intervention to college students.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be de-identified both by removing identifying information and any other procedures necessary to keep the data from being re-identified using known methods. The independent and dependent variables relevant to the primary outcomes will be shared
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon submission of the manuscript to a peer-reviewed journal (Anticipated date: 8-1-2020). The data will be available open access thereafter.
Access Criteria: The de-identified data will be shared open access

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT04082052/SAP_000.pdf